CLINICAL TRIAL: NCT01020630
Title: A Randomized, Placebo-controlled Phase II Trial Investigating SUNITINIB Versus Placebo in Patients With Chemorefractory Advanced Adenocarcinoma of the Stomach or Lower Esophagus Treated With Chemotherapy FOLFIRI
Brief Title: Sunitinib in Patients With Advanced Gastric Cancer and Treated With FOLFIRI
Acronym: SUN-CASE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: PD Dr Markus Möhler (Other)
Responsible Party: Sponsor-Investigator, PD Dr Markus Möhler, PD Dr., Johannes Gutenberg University Mainz
Organization: Johannes Gutenberg University Mainz (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2009-02-SUN-Case
Record Dates: First submitted 2009-11-23; First posted 2009-11-25 (Estimated); Last update posted 2014-05-14 (Estimated); Status verified 2014-05

CONDITIONS: Adenocarcinoma
Keywords: adenocarcinoma of stomach; adenocarcinoma of lower oesophagus; sunitinib; FOLFIRI
MeSH Terms: conditions — Adenocarcinoma | interventions — Sunitinib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sunitinib (Experimental): 25 mg (2 capsules of 12.5 mg) for oral administration
  Interventions: Drug: Sunitinib
- Placebo (Placebo Comparator): 2 capsules for oral administration
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Sunitinib — Sunitinib will be orally administered at 25 mg once daily (in the morning without regards to meals) for 4 consecutive weeks followed by a 2-week rest period to comprise a complete cycle of 6 weeks.
  Other Names: Sutent
  Arms: Sunitinib
Drug: Placebo — Placebo will be orally administered once daily (in the morning without regards to meals) for 4 consecutive weeks followed by a 2-week rest period to comprise a complete cycle of 6 weeks.
  Arms: Placebo

SUMMARY:
This trial will be conducted to evaluate the efficacy, safety and tolerability of SUNITINIB as add-on therapy with a widely used second-line palliative FOLFIRI chemotherapy in patients with chemo-refractory advanced or metastatic adenocarcinoma of stomach or lower esophagus (mGC).

There is a clear scientific rationale for the use of Sunitinib to treat patients with mGC. Despite recent therapeutic advances, the median overall survival (OS) in patients with mG is still ≤ 12 months. Therefore, newer agents with novel mechanisms of action are desperately needed for treatment of these patients.

DETAILED DESCRIPTION:
In parallel to the efforts in front-line therapy, second-line protocols like irinotecan-based regimens have been established in clinical trials for those patients. As many patients are still in good performance status and present with low tumor burden after failure of first-line chemotherapy, they clearly benefit from second-line treatment.

Sunitinib inhibits the receptor tyrosine kinases (RTKs) involved in tumor proliferation and angiogenesis, specifically the VEGFR, PDGFR, KIT, FLT-3, and RET. The VEGF pathway has been shown to be a significant factor in metastatic gastric cancer.

The safety and efficacy of Sunitinib as single agent for the treatment of mGC has been determined and support the proposed clinical study with FOLFIRI in combination with Sunitinib in the treatment of patients with mGC.

Patients included in this trial suffer from advanced or metastatic adenocarcinoma of stomach or lower esophagus. They have failed to respond at least to one standard palliative first-line therapy (based on docetaxel and/or cisplatin plus 5-FU). Irinotecan/FA/5-FU can be determined as one established second-line treatment to be available for these patients.

Taken together, treatment of those patients with Sunitinib combined with standard chemotherapy FOLFIRI offers the chance to benefit from a new innovative therapy with acceptable side effects.

ELIGIBILITY:
Inclusion Criteria:

* Signed and dated informed consent before the start of specific protocol procedures
* Histological proven gastric adenocarcinoma including adenocarcinoma of the esophagogastric junction or lower esophagus
* Failure of any prior chemotherapy (docetaxel and/or platinum-based chemotherapy); but patient has not previously received FOLFIRI treatment
* Measurable metastatic disease according to the RECIST criteria patients aged 18 years and older
* karnofsky index 100 - 70 %
* Life expectancy > 12 weeks
* Adequate hematological, hepatic and renal functions
* At least 3 weeks from previous docetaxel- and/or platinum-based chemotherapy
* Recovery from hematological side effects (CTC grade <1) and non-hematological side effects (CTC grade=<1) of any prior therapy (except oxaliplatine induced neuropathy CTC grade =<2)

Exclusion Criteria:

* History of another primary malignancy >3 years, with the exception of non-melanoma skin cancer and in situ carcinoma of the uterine cervix
* Any prior palliative radiotherapy of the target lesions
* Concurrent treatment with any other medicinal anti-cancer therapy
* Prior treatment with a VEGF, VEGFR or RTK inhibitor, or prior enrolment on this study
* Known allergic/hypersensitivity reaction to any of the components of the treatment
* Treatment with potent CYP3A4 inhibitor within 7 days of Sunitinib/placebo dosing or with potent CYP3A4 inducer within 12 days of Sunitinib/placebo dosing
* Other serious illness or medical conditions within the last 12 months prior to study drug administration: Unstable cardiac disease despite treatment; myocardial infarction within 12 months prior to study entry; congestive heart failure NYHA grade 3 and 4; Hypertension that cannot be controlled by medication ; ongoing cardiac dysrhythmias of NCI CTCAE grade >2, atrial fibrillation of any grade, or QTc interval >450 msec for males or >470 msec for females; History of significant neurologic or psychiatric disorders including dementia or seizures; Active uncontrolled infection; History of clinically significant bleeding within the past 6 months, including hemoptysis or haematuria, or underlying coagulopathy; Active disseminated intravascular coagulation; Cerebrovascular accident including transient ischemic attack; Pulmonary embolus; Bowel obstruction or chronic diarrhoea, history or presence of inflammatory enteropathy or extensive intestinal resection; History of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within 6 months prior to study enrolment, unless affected area has been removed surgically
* Known deficit in DPD
* Hypercalcemia not controlled by bisphosphonates
* Contraindications to the use of atropine
* Pregnant or lactating women; female patients who are pregnant or lactating or men and women of reproductive potential not willing or not able to employ an effective method of birth control/contraception to prevent pregnancy during treatment and for 3 months after discontinuing study treatment
* Known drug abuse/alcohol abuse
* Current, recent, or planned participation in an experimental treatment drug study other than this protocol
* Major surgical procedure, open biopsy or significant traumatic injury within 4 weeks before starting treatment; anticipation of need for major surgical procedure (e.g. impending bowel obstruction) during the course of the study
* History of other medical or psychiatric condition, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug or that might affect the interpretation of the results of the study or render the patient at high risk from treatment complications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2009-11; Primary Completion 2012-11 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
The primary endpoint is the Progression-free survival (PFS) according to RECIST V1.1. | Average time period: up to one year (participants are followed until progression or death)

SECONDARY OUTCOMES:
Objective response rate (CR + PR) according to RECIST | Average time period: up to one year (participants are followed until progression or death)
Safety and tolerability | one year

CONTACTS AND LOCATIONS:
Overall Officials: Markus Moehler, MD, Principal Investigator — Johannes Gutenberg University Mainz, 1. Med. Klinik
Locations (16):
- Germany (16):
  - Krankenhaus Nordwest, Frankfurt, Germany
  - Universitätsmedizin Mainz, 1. Med. Klinik, Mainz, Rhineland-Palatinate
  - Gesundheitszentrum St. Marien, Amberg
  - Helios Klinikum Berlin-Buch, Berlin
  - Universitätsmedizin Berlin Charite, Berlin
  - Evangelisches Krankenhaus Bielefeld, Bielefeld
  - Universitätsklinikum Essen, Essen
  - Kliniken Essen-Mitte, Essen
  - Martin-Luther-Universität Halle-Wittenberg, Halle
  - MVZ für Innere Medizin in Hamburg-Eppendorf, Hamburg
  - Universitätsklinikum des Saarlandes, Homburg
  - Klinikum Ludwigsburg Medizinische Klinik I, Ludwigsburg
  - Technische Universität München, München
  - Universitätsklinikum Rostock Klinik für Innere Medizin, Rostock
  - Leopoldina-Krankenhaus der Stadt Schweinfurt gGmbH, Schweinfurt
  - Klinikum Weiden, Weiden

REFERENCES:
- [Derived] Moehler M, Gepfner-Tuma I, Maderer A, Thuss-Patience PC, Ruessel J, Hegewisch-Becker S, Wilke H, Al-Batran SE, Rafiyan MR, Weissinger F, Schmoll HJ, Kullmann F, von Weikersthal LF, Siveke JT, Weusmann J, Kanzler S, Schimanski CC, Otte M, Schollenberger L, Koenig J, Galle PR. Sunitinib added to FOLFIRI versus FOLFIRI in patients with chemorefractory advanced adenocarcinoma of the stomach or lower esophagus: a randomized, placebo-controlled phase II AIO trial with serum biomarker program. BMC Cancer. 2016 Aug 31;16(1):699. doi: 10.1186/s12885-016-2736-9. PMID 27582078